CLINICAL TRIAL: NCT04271254
Title: Quantitative PET-MRI Imaging Correlated With Transcriptome Analysis for Noninvasive Characterization of Renal Cell Carcinomas
Brief Title: PET/MR Characterization of Renal Cell Carcinomas
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding insufficiency.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC 1930
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Results first posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PET/MR (Experimental): Each patient will undergo one combined PET/MR scan prior to surgery. The PET/MR scans are for research purposes and not part of the patient's standard of care.
  Interventions: Diagnostic Test: PET/MR

INTERVENTIONS:
Diagnostic Test: PET/MR — Patient will be scheduled for a pre-surgery PET/MR within four weeks of scheduled surgery.

SUMMARY:
Purpose: To evaluate the utility of simultaneous positron emission tomography (PET) and magnetic resonance imaging (MRI) in characterizing the molecular subtypes of clear cell renal cell carcinomas (ccRCC) to potentially inform prognosis and treatment decisions.

Participants: Seventeen subjects diagnosed with clear-cell renal cell carcinoma (ccRCC) will be imaged in a single session on PET-MRI.

Procedures (methods): The investigators will image 17 ccRCC subjects on simultaneous PET-MRI and quantify the metabolically-active fraction of the tumor from images. Ten core samples will be taken from each tumor post-surgery and classified as ccA or ccB subtype using transcriptome analysis. The imaging-based measures will be correlated with the fraction of tumor cores classified as ccB.

DETAILED DESCRIPTION:
Simultaneous PET/MR imaging [1]-[7] offers exciting opportunities to visualize and quantify soft-tissue tumors [2]. MRI offers superb soft-tissue contrast for anatomical information as well as a flexible suite of other techniques providing functional and physiological information. PET offers sensitive molecular imaging via radioactive tracers and is widely used for assessment of tumor glucose metabolism. Together, the two modalities provide complementary, synergistic information. Because of MRI's superior soft-tissue contrast, it is considered a much better anatomical guide for PET quantitative analyses for tumors in soft tissue regions as compared to standard-of-care PET-CT. Simultaneous PET-MR also provides inherently-aligned PET and MR, efficient simultaneous acquisition, and the opportunity for new approaches to PET quantitative analysis guided by detailed MR images.

Nonmetastatic clear cell renal cell carcinomas are generally treated with nephrectomy, although research has subclassified them into two [8] or as many as four [9] subtypes based on gene expression; the subtypes have been shown to have differing prognoses and progression [8]-[11]. The investigators focus primarily on the two subtypes ccA and ccB [8] and ask whether these two exhibit distinct PET-MRI imaging characteristics that can be used to subtype them noninvasively. An eight-subject pilot study conducted on PET-MRI at UNC demonstrated that quantitative PET-MRI imaging, using nonstandard measures incorporating the entire tumor, was strongly correlated with presence or absence of ccB patterns in the tumors [12]. Transcriptome analysis results from the study justified the import of PET in noting that many of the upregulated genes associated with ccB were involved in glucose transport and metabolism, the mediators of 18-FDG uptake. Thus, there is a strong biologic rationale as to why PET-MRI could predict ccB burden, but the small number of subjects in that study limits confidence.

Also, the fact that these tumors are highly heterogeneous suggests that imaging alone provides an opportunity for early characterization of ccB burden across the entire tumor where gene expression profiling would be invasive and costly. Also, with the excellent soft-tissue contrast of MRI, the system has the potential for greater anatomical detail to guide interpretation of FDG activity. UNC has one of the few PET-MR scanners in the country, making it one of few centers in the US capable of conducting this study.

This is a prospective study of the use of combined PET-MR [1-7] for prediction of tumor subtype composition in ccRCC. Additional data analysis using the prior study from UNC suggests a strong correlation between the fraction of the tumor exhibiting moderate to high FDG uptake and the number of cores found to be ccB type. These results guide the hypothesis of this study: the metabolically-active tumor volume fraction derived from simultaneous PET-MRI imaging of clear-cell renal cell carcinomas is correlated with the fraction of tumor cores classified as ccB subtype from transcriptome analysis. If so, in the future, application of PET-MRI may offer prognostic information and opportunities for risk stratification.

ELIGIBILITY:
Inclusion Criteria:

1. Age ? 18 years of age (no upper age limit)
2. Signed, IRB-approved written informed consent
3. Must have clinically-suspected ccRCC based on prior imaging with tumor size >= 7 cm.
4. Planned nephrectomy schedule that can accommodate a MR-FDG-PET scan within 4 weeks prior to surgery.
5. Must be able to meet size restrictions for the PET-MR scanner.
6. Must be able to understand and comply with study procedures for the entire length of the study.
7. Must receive their nephrectomy at UNC Hospitals.
8. If patient has a history of prior malignancy, including melanoma, patient must be cancer-free for three or more years. Non-melanoma skin cancers will be included even if not cancer-free for three years.
9. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to PET/MRI.

Exclusion Criteria:

1. Inability to tolerate MRI (e.g., inability to lie flat for >1 hour)
2. Presence of pacemaker, intracranial aneurysm clip, bladder stimulator, cochlear implant or metal near eyes or near pelvis that would create excessive imaging artifact
3. Failure of two blood glucose tests (blood glucose level greater than 200 mg/dL) on day of first scheduled scan visit and on rescheduled day.
4. Body Mass Index (BMI) > 35
5. Patient receiving neoadjuvant therapy for RCC
6. Pregnancy or lactating female
7. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study
8. Evidence of distant disease on physical exam or initial imaging
9. Medical conditions precluding chemotherapy or curative intent surgery
10. Incarcerated or otherwise institutionalized at time of enrollment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Lalush, Principal Investigator — UNC Biomedical Engineering
Locations (1):
- UNC- Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 08/01/2020- 06/14/2023, 5 subjects consented and enrolled in the study at one center in North Carolina.
Pre-assignment Details: although 5 subjects signed the consent and enrolled in the study, 2 subjects underwent Positron Emission Tomography (PET) and magnetic resonance (MR) imaging and have available tissue specimens. The tumor type was not renal cell carcinoma in one out of 2 subjects with tissue specimens. Only 1 subject has an available tissue specimen.
Groups:
- PET/MR: Each patient will undergo one combined PET/MR scan prior to surgery. The PET/MR scans are for research purposes and not part of the patient's standard of care.
  PET/MR: The patient will be scheduled for a pre-surgery PET/MR within four weeks of the scheduled surgery.
Period: Overall Study
Arm/Group | PET/MR
Started | 5
Completed | 2
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | PET/MR
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between PET Activity Distribution and Tumor Subtype Composition
Description: The correlation between Positron Emission Tomography (PET) activity distribution and tumor subtype composition will be assessed as the relation of PET activity estimates (in the form of fractional tumor volume over PET SUV threshold of 2.0) and the fraction of tumor cores classified as ccB subtype by transcriptome analysis. Ten core samples will be taken from each tumor at surgery time and will be examined with a panel of 34 genes found to distinguish ccA and ccB subtypes.
  The single subject's tissue analysis will not done immediately following surgery because the study was planned from the beginning to bank the tissue samples and analyze them all at once at the completion of the study.
Time Frame: PET/MR scans will be taken within four weeks prior to surgery. Tissue samples will be taken at the time of surgery. (from the PET/MR scan to Surgery Day=Day 1)
Population: Data was not collected. The study was close to accrual before reaching target accrual because the internal funding source for the study recommended closure due to poor accrual. Only one subject meeting the study criteria completed the imaging portion of the study and has a tissue sample for transcriptome analysis. Transcript analysis was not performed for a single subject since the result of a single subject would not provide a conclusion.
Arm/Group | PET/MR
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 -Until Day 2 (Positron Emission Tomography/ Magnetic Resonance scan was performed, approximately 4 weeks before surgery
Groups:
- PET/MR: Each patient will undergo one combined PET/MR scan prior to surgery. The PET/MR scans are for research purposes and not part of the patient's standard of care.
  PET/MR: The patient will be scheduled for a pre-surgery PET/MR within four weeks of the scheduled surgery.
  The subjects who underwent PET/MR were included in the Adverse Event evaluation.
Arm/Group | PET/MR
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT04271254/Prot_SAP_000.pdf